CLINICAL TRIAL: NCT00381524
Title: Special Projects of National Significance
Brief Title: HIV Prevention in the Primary Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Edward Hook III, MD, Professor of Medicine, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: F040223020; 6 H97HA01191-03-02 (HRSA)
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2009-11

CONDITIONS: Human Immunodeficiency Virus
Keywords: human immunodeficiency virus; behavior change
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

INTERVENTIONS:
Behavioral: Increase condom use — Voluntary increase in condom use

SUMMARY:
In the third decade of the HIV pandemic, what was once a uniformly and rapidly fatal disease has been transformed into a chronic illness by advances in the understanding of HIV pathogenesis and therapeutics. As a result, HIV-infected individuals are living longer and better lives. This phenomenon, coupled with a continued steady rate of new HIV infections in this country, has led to the highest U.S. HIV prevalence rates since the beginning of the epidemic. In the past, HIV prevention efforts were separate from routine primary care delivery due to multiple factors including stigma and time constraints. Recent events, including increases in sexually transmitted disease (STD) rates among HIV-infected persons and evidence that infected individuals can be super-infected by HIV strains resistant to antiretroviral therapy, have inspired the SPNS program initiative to develop demonstration projects for interventions to reduce risky sexual exposures among HIV-infected patients receiving primary care.

DETAILED DESCRIPTION:
Goals of the Demonstration Project. The goals of this project are as follows:

Goal 1: To utilize recent technological advances and refine a theory-based, computerized intervention system currently being evaluated in a Birmingham STD clinic. Our proposed interventions will target men-who-have-sex-with-men (MSM) and will be designed to: increase condom use for specific sexual activities with both main and casual (other) partners; decrease numbers of sexual partners among those reporting multiple partners; and increase the frequency of HIV serostatus disclosure to sexual partners.

Goal 2: To evaluate a computer-guided, theory-based, provider-delivered intervention in the context of standard care in an HIV primary care facility in collaboration with the Center for AIDS Prevention Studies (CAPS). We will test the following hypotheses after 18 months of follow-up:

Hypothesis 1: That the proportion of HIV-positive MSM reporting 100% condom use with main partners will be significantly increased in the intervention group compared to the usual care group.

Hypothesis 2: That the proportion of patients reporting 100% condom use with casual partners will be significantly increased among patients in the intervention group compared to the usual care group.

Hypothesis 3: That the proportion of patients with multiple sexual partners will be significantly reduced among intervention group participants compared with the usual care group.

Hypothesis 4: That the proportion of HIV-positive MSM who disclose their HIV status to sex partners who are HIV-negative or are of unknown HIV status will be significantly increased among the patients receiving the intervention compared to the patients in the usual care group.

Goal 3: In collaboration with the Center and SPNS program, to conduct a holistic evaluation of the intervention program.

Goal 4: To compare the cumulative incidence of symptomatic and asymptomatic treatable STDs (gonococcal and chlamydial infections) between patients in the intervention and usual care groups.

ELIGIBILITY:
Inclusion Criteria:

* Active male patients over the age of 16 receiving routine primary care at the 1917 Clinic, reporting sexual contact with another man in the previous 6 months. Active patients will be defined as new patients (patients' first visit) with plans to continue follow-up at 1917 Clinic or an established patient seen at least once during the past year
* Willingness to follow-up for at least 18 months
* Ability to sign informed consent.

Exclusion Criteria:

* Female patient
* Male patient who is unwilling to follow-up for at least 18 months
* Male patient who is not a primary care patient at the clinic
* Unwillingness or inability to sign informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2004-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Proportion of participants reporting 100% condom use preintervention versus post intervention | End of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Edward W Hook, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB 1917 Clinic, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No